CLINICAL TRIAL: NCT04523987
Title: A Pilot Study of Ciprofloxacin Plus Gemcitabine and Nab-Paclitaxel Chemotherapy in Patients With Metastatic Pancreatic Ductal Adenocarcinoma.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA02/07/18
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Ciprofloxacin; Gemcitabine; Nab-Paclitaxel Chemotherapy
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: This is a single-center, pilot study evaluating the addition of Ciprofloxacin (study drug) to standard-of-care gemcitabine and nab-paclitaxel chemotherapy in treatment-naïve metastatic PDAC patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- gemcitabine and nab-paclitaxel chemotherapy (Experimental): Patients who are recommended gemcitabine and nab-paclitaxel chemotherapy as a standard-of-care by their treating physician will be offered to participate in this study.
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Subjects enrolled will be administered oral ciprofloxacin twice a day throughout the course of each 28-day cycle of gemcitabine and nab-paclitaxel chemotherapy.

SUMMARY:
This is a single-center, pilot study evaluating the addition of Ciprofloxacin (study drug) to standard-of-care gemcitabine and nab-paclitaxel chemotherapy in treatment-naïve metastatic PDAC patients. Patients who are recommended gemcitabine and nab-paclitaxel chemotherapy as a standard-of-care by their treating physician will be offered to participate in this study.

DETAILED DESCRIPTION:
Oral ciprofloxacin (study drug) will be administered twice a day throughout each 28-day cycle of gemcitabine and nab-paclitaxel chemotherapy. The patient will start taking ciprofloxacin from the evening of day 1 of chemotherapy and end on the morning of day 29 of each cycle.

Ciprofloxacin tablets should be taken in the morning and evening at about the same time each day. Swallow the tablet whole. Do not split, crush or chew the tablet. Ciprofloxacin can be taken with or without food

With each study visit, the physician will prescribe 1-month supply of oral ciprofloxacin to be taken home and self-administered by the patient. The physician will have to indicate "pancreatic cancer microbiome study" on the remarks column for each cycle oral ciprofloxacin is ordered.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent. Written informed consent must be obtained prior to performing any study-related procedures.
* Age ≥ 21 years
* Histologically or cytologically confirmed, treatment-naïve, locally advanced or metastatic pancreatic adenocarcinoma planned to commence on gemcitabine and nab-paclitaxel chemotherapy.
* Patient must have measurable disease as defined by the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1 guidelines)
* Life expectancy >3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* CrCl ≥ 30 ml/min

Exclusion Criteria:

* Known hypersensitivity or allergy to ciprofloxacin or other quinolones
* On tizanidine or theophylline and unable to stop these medication
* Known QTc prolongation (QTc >500 msec) or torsade de pointes
* Presence of Clostridium difficile-associated diarrhea or colitis
* Known history of myasthenia gravis
* Known G6PD deficiency

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Antitumor Effect - Solid Tumors | 4 years
  Patients are be re-evaluated for response every 8-12 weeks (±10 days), per standard-of-care.
  Response and progression will be evaluated in this study using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Ean Chee, Principal Investigator — cheng_ean_chee@nuhs.edu.sg
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Ertz-Archambault N, Keim P, Von Hoff D. Microbiome and pancreatic cancer: A comprehensive topic review of literature. World J Gastroenterol. 2017 Mar 14;23(10):1899-1908. doi: 10.3748/wjg.v23.i10.1899. PMID 28348497
- [Background] Farrell JJ, Zhang L, Zhou H, Chia D, Elashoff D, Akin D, Paster BJ, Joshipura K, Wong DT. Variations of oral microbiota are associated with pancreatic diseases including pancreatic cancer. Gut. 2012 Apr;61(4):582-8. doi: 10.1136/gutjnl-2011-300784. Epub 2011 Oct 12. PMID 21994333